CLINICAL TRIAL: NCT01369615
Title: An Open-label, Extension Study to Assess the Long-Term Safety of Twice Daily Oxycodone Hydrochloride Controlled-release Tablets in Opioid Experienced Children Who Completed the OTR3001 Study
Brief Title: Long-Term Safety of Twice Daily Oxycodone Hydrochloride Controlled-release Tablets in Children Who Completed OTR3001
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OTR3002; 2011-002235-26 (EudraCT Number)
Record Dates: First submitted 2011-06-07; First posted 2011-06-09 (Estimated); Results first posted 2015-01-15 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-08

CONDITIONS: Pain
Keywords: Malignant pain; Nonmalignant pain; Pain; Pediatric; Opioid; Moderate to severe
MeSH Terms: conditions — Pain | interventions — Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oxycodone HCl controlled-release (Experimental): Oxycodone hydrochloride controlled-release tablets
  Interventions: Drug: Oxycodone hydrochloride controlled-release tablets

INTERVENTIONS:
Drug: Oxycodone hydrochloride controlled-release tablets — Oxycodone hydrochloride controlled-release tablets at strengths of 10, 15, 20, 30, or 40 mg (20 mg to 240 mg daily) every 12 hours.
  Other Names: OxyContin

SUMMARY:
The purpose of this study is to characterize the long-term safety of oxycodone hydrochloride (HCl) controlled-release (CR) tablets in opioid experienced pediatric patients aged 6 to 17 years, inclusive, with moderate to severe malignant and/or nonmalignant pain requiring opioid therapy who completed the 4 -week treatment period in OTR3001.

ELIGIBILITY:
Inclusion Criteria include:

1. Male and female patients aged 6 to 17 years, inclusive, who completed the 4-week study drug treatment in study OTR3001 and who, based on the investigator's judgment, will benefit from continuing treatment with oxycodone HCl CR 20 to 240 mg/day for the management of moderate to severe malignant or nonmalignant pain;
2. Patients must have tolerated the oxycodone HCl CR therapy in OTR3001 as demonstrated at the start of the study;
3. Patients must be willing and able to swallow the oxycodone HCl CR tablets whole.

Exclusion Criteria include:

1. Patients with ongoing adverse events in OTR3001 that, in the investigator's opinion, disqualify them from participation in the study;
2. Female patients who are pregnant or lactating;
3. Patients requiring opioid at doses equivalent to < 20 mg/day or > 240 mg/day oxycodone for treatment of their malignant or nonmalignant pain;
4. Patients who are allergic to oxycodone or have a history of allergies to other opioids (this criterion does not include patients who have experienced common opioid side effects [eg, nausea, constipation]);
5. Patients who are contraindicated for the use of opioids;
6. Patients who are currently being maintained on methadone for pain;
7. Patients who have an abnormality on vital signs, physical examination, or laboratory testing significant enough that the investigator deems the patient is not appropriate for the study;
8. Patients who have any planned surgery during the course of the study, with the exception of the placement of central or peripheral venous access devices;
9. Patients currently taking an investigational medication/therapy other than the study drug (oxycodone HCl CR) at the start of screening or during the study.

Other protocol specific inclusion/exclusion criteria may apply.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2011-10; Primary Completion 2013-12 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (13):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Bayview Research Group, LLC, Paramount, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Jackson Memorial Hospital, Miami, Florida
  - University of Kentucky, Lexington, Kentucky
  - Mercy Clinic Children's Cancer and Hematology Center, St Louis, Missouri
  - New York University Langone Medical Center, New York, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Presbyterian Blume Pediatric Hematology & Oncology Clinic, Charlotte, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - The Children's Hospital at Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Children's Medical Center of Dallas, Dallas, Texas
- Schneider Children Medical Center of Israel, Petah Tikva, Israel

REFERENCES:
- See also: Product Information — http://www.purduepharma.com/wp-content/uploads/2015/08/302940-0G-August-2015.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient First Visit: 05-January-2012; Last Patient Last Visit: 09-December-2013. The study was conducted at 14 medical/research sites in the United States and Israel.
Pre-assignment Details: Opioid-experienced pediatric patients with moderate to severe malignant and/or nonmalignant pain requiring around-the-clock opioid therapy were eligible for open-label Extension Study OTR3002 if they completed the 4-week treatment period Core Study OTR3001 and could benefit from continued treatment with oxycodone HCl CR 20 to 240 mg total daily.
Groups:
- 6 to < 12 Years: Children 6 to < 12 years of age
- ≥ 12 to ≤ 16 Years: Although the protocol for study OTR3002 defined the age range as 6 to 17 years inclusive, no patients greater than 16 years of age were included in the study. Therefore the data summaries presented the upper limit of the older age group as ≤ 16 years.
Period: Overall Study
Arm/Group | 6 to < 12 Years | ≥ 12 to ≤ 16 Years
Started | 9 | 14
Completed | 9 | 12
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: The extension safety population was the group of patients who received at least 1 dose of study drug during the Extension Study.
Groups:
- ≥ 12 to ≤ 16 Years: Children 12 to ≤ 16 years of age
- Total: Total of all reporting groups
Arm/Group | 6 to < 12 Years | ≥ 12 to ≤ 16 Years | Total
Number analyzed (Participants) | 9 | 14 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.9 (1.76) | 14.3 (1.49) | 12.6 (2.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 3 | 7 | 10
Race/Ethnicity, Customized [Number; unit: participants]
  White | 6 | 10 | 16
  Black or African American | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Adverse Events as a Measure of Safety.
Description: Safety assessments included adverse events (AEs), vital sign measurements, clinical laboratory test results, and somnolence (University of Michigan Sedation Scale [UMSS]). Safety variables were summarized descriptively within age group for the extension safety population.
Time Frame: Up to 6 months (during the study) and 7-10 days poststudy (safety follow-up assessment).
Population: as for baseline characteristics
Measure: Number; unit: participants
Groups:
- 6 to < 12 Years; ≥ 12 to ≤ 16 Years: Test treatment: open-label oxycodone HCl CR tablets, 20 mg to 240 mg total daily
Arm/Group | 6 to < 12 Years | ≥ 12 to ≤ 16 Years
Number analyzed (Participants) | 9 | 14
participants
  Serious adverse events | 3 | 2
  All other adverse events in ≥ 5% of patients | 8 | 8

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were reported from start of study participation through the period beyond study completion.
Description: AEs were learned of through spontaneous reports and/or patient interview, or were observed during physical examinations or other safety assessments. Ongoing AEs were followed until resolution or 30 days after last study drug dose. Serious AEs up to 30 days following the last study visit were followed until the AE or sequelae resolved or stabilized.
Groups:
- ≥ 12 to ≤ 16 Years: Children ≥ 12 to ≤ 16 years of age
Arm/Group | 6 to < 12 Years | ≥ 12 to ≤ 16 Years
Serious Adverse Events (participants affected / at risk) | 3/9 | 2/14
Other Adverse Events (participants affected / at risk) | 8/9 | 8/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 6 to < 12 Years (N=9) | ≥ 12 to ≤ 16 Years (N=14)
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 6 to < 12 Years (N=9) | ≥ 12 to ≤ 16 Years (N=14)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 0 | 1
Auricular swelling (Ear and labyrinth disorders) | 0 | 1
External ear pain (Ear and labyrinth disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0
Eye pain (Eye disorders) | 1 | 0
Mydriasis (Eye disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 2
Adverse drug reaction (General disorders) | 0 | 1
Cyst (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Inflammation (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Vaginal infection (Infections and infestations) | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 1
Platelet count decreased (Investigations) | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Blood magnesium decreased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1
Oxygen saturation decreased (Investigations) | 1 | 0
Respiratory rate (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Sedation (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Scar (Skin and subcutaneous tissue disorders) | 1 | 0
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Scar excision (Surgical and medical procedures) | 0 | 1
Flushing (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Enrollment for study OTR3002 was closed by Purdue Pharma L.P. on 01-January-2014 due to administrative reasons not related to safety.

Interpretation is limited by the small number of patients in each age group in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days